CLINICAL TRIAL: NCT02651454
Title: A Pilot Study Exploring the Efficacy and Safety of Herbal Medicine on Korean Obese Women With Metabolic Syndrome Risk Factors - Double Blinded, Randomized, Multicenter, Placebo Controlled Clinical Trial -
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Gachon University Gil Oriental Medical Hospital (Other)
Collaborators: Sangji University Oriental Medical Hospital, Korea (Unknown); DongGuk University (Other)
Responsible Party: Principal Investigator, Yun-Kyung Song, KMD, PhD, Gachon University Gil Oriental Medical Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ISEE_2015_OBESITY
Record Dates: First submitted 2016-01-05; First posted 2016-01-11 (Estimated); Last update posted 2021-04-12 (Actual); Status verified 2021-04

CONDITIONS: Metabolic Syndrome; Obesity
Keywords: metabolic syndrome; Daesiho-tang; Taeeumjowi-tang; Korean medicine
MeSH Terms: conditions — Metabolic Syndrome; Obesity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Daesiho-tang (Experimental): Dose: 6g, three times a day, each taken before or between meals for 12 weeks
  Interventions: Drug: Daesiho-tang
- Jowiseungcheung-tang (Experimental): Dose: 6g, three times a day, each taken before or between meals for 12 weeks
  Interventions: Drug: Chowiseungcheng-tang
- Placebo (Placebo Comparator): Dose: 6g, three times a day, each taken before or between meals for 12 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Daesiho-tang — Usage: 6g, three times a day, each taken before or between meals for 12 weeks Manufacturing company: HANPOONG PHARM & FOODS Co. Ltd.
  Other Names: DSHT; Elsion Granule
  Arms: Daesiho-tang
Drug: Chowiseungcheng-tang — Usage: 6g, three times a day, each taken before or between meals for 12 weeks Manufacturing company: Hanzung Pharmaceutical. co. Ltd.
  Other Names: CST
  Arms: Jowiseungcheung-tang
Drug: Placebo — Usage: 6g, three times a day, each taken before or between meals for 12 weeks Manufacturing company: HANPOONG PHARM & FOODS Co. Ltd.
  Arms: Placebo

SUMMARY:
The Purpose of this trial is to investigate the efficacy and safety of Daesiho-tang and Taeeumjowi-tang on Korean obese Women with metabolic syndrome Risk factors

ELIGIBILITY:
Inclusion Criteria:

* Female aged 18 to 65 years
* Subject must included at least one or more of the following symptoms below

  * BMI of 30 kg/㎡ or more;
  * BMI between 25 and 29.9kg/㎡ with hypertension, taking medication or SBP ≥ 140mmHg or DBP ≥ 90mmHg at the screening visit
  * BMI between 25 and 29.9kg/㎡ with non-insulin-dependent diabetes mellitus, taking medication or fasting blood glucose > 126mg/dL at the screening visit
  * BMI between 25 and 29.9kg/㎡ with hyperlipidemia, taking medication or total cholesterol ≥ 200mg/dL or Triglyceride ≥ 150mg/dL at screening visit
* Agreed to low-calorie diet during the trial
* Written informed consent of the trial

Exclusion Criteria:

* Endocrine diseases associated with weight gain, such as hypothyroidism, Cushing's syndrome, etc.
* Heart disease (heart failure, angina pectoris, myocardial infarction)
* Cholelithiasis
* Severe renal disability (SCr > 2.0 mg/dL)
* Severe liver disability (2.5 fold of normal high range value on Alanine Aminotransferase [ALT], Aspartate Aminotransferase [AST], alkaline phosphatase)
* History of narrow angle glaucoma
* History of stroke or temporary ischemic cardioplegia
* History of eating disorder such as anorexia nervosa or bulimia nervosa, etc.
* Use of medication that can affect on weight within last 3 months (appetite suppressant, laxative, oral steroid, thyroid hormone, amphetamine, cyproheptadine, phenothiazine or medications can affect on absorption, metabolism, excretion)
* Use of CNS stimulant medication for weight loss
* Forbidden treatment (Insulin, hypoglycemic agent, antidepressant, antiserotonin agent, barbiturate, antipsychotic, medication concerns of abuse)
* history of weight loss surgery, such as bariatric surgery, etc.
* Subjects who are judged to be inappropriate for the clinical study by the researchers
* Women who were pregnant, lactating or have the chances of pregnancy who do not agree to proper contraception (birth-control pill, hormone implant, IUD, spermicide, condom, abstinence, etc.)
* Use of other investigational product within last 1 month
* 10 percent reduction in body weight over 6 months
* Decided to quit smoking over the last 3 months or have irregular smoking habits

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2015-12-31 (Actual); Primary Completion 2020-05-02 (Actual); Study Completion 2020-12-02 (Actual)

PRIMARY OUTCOMES:
Changes from baseline in body weight | baseline, 12 weeks

SECONDARY OUTCOMES:
Changes from baseline in body fat percentage | baseline, 4,8,12,16 weeks
Changes from baseline in fat mass | baseline, 4,8,12,16 weeks
Changes from baseline in Waist circumference | baseline, 4,8,12,16 weeks
Changes from baseline in Waist/hip ratio | baseline, 4,8,12,16 weeks
Changes from baseline in Body mass index | baseline, 4,8,12,16 weeks
Changes from baseline in Lipid profile | Screening visit, 12 weeks
Changes from baseline in C-reactive protein (CRP) | Screening visit, 12 weeks
Changes from baseline in blood glucose | Screening visit, 12 weeks
Changes from baseline in abdominal visceral fat area | baseline, 12 weeks
Korean Obesity-related Quality of Life (QoL) scale | baseline, 12 weeks
Korean version of Eating Attitudes Test-26 | baseline, 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Yun-Kyung Song, KMD, Principal Investigator — Gachon University Gil Oriental Medical Hospital
Locations (1):
- Gachon University Gil Oriental Medical Hospital, Incheon, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kim HJ, Ko Y, Kim H, Cha YY, Jang BH, Song YK, Ko SG. A pilot study exploring the efficacy and safety of herbal medicine on Korean obese women with metabolic syndrome risk factors: Double blinded, randomized, multicenter, placebo controlled study protocol clinical trial. Medicine (Baltimore). 2020 Jan;99(5):e18955. doi: 10.1097/MD.0000000000018955. PMID 32000419